CLINICAL TRIAL: NCT04330183
Title: Low Dose Ketamine for Acute Pain Crisis in Patients With Sickle Cell Disease
Brief Title: Low Dose Ketamine and Acute Pain Crisis
Acronym: LDK-SCD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1481617
Record Dates: First submitted 2020-03-23; First posted 2020-04-01 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Sickle Cell Crisis
Keywords: ketamine; emergency department; acute pain crisis
MeSH Terms: conditions — Vaso-Occlusive Crises; Emergencies | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Normal Saline (Placebo Comparator): Patients here will be administered 3cc of normal saline as placebo
  Interventions: Drug: Normal Saline
- Ketamine Interventions (Experimental): Patients will be administered weight based 0.3mg/kg of ketamine
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — 0.3mg/kg of ketamine
  Arms: Ketamine Interventions
Drug: Normal Saline — 3cc of normal saline
  Arms: Normal Saline

SUMMARY:
BACKGROUND:

Current treatment standard for acute pain crisis in sickle cell disease (SCD) is largely supportive care: opioid analgesics, hydration, oxygen, and blood transfusion. Sickle cell disease (SCD) is a chronic condition associated with serious and disabling acute consequences such as a vaso-occlusive (VOC) or pain crisis. Uncontrolled pain is the hallmark of a VOC, and often results in acute unscheduled care in the patient's clinic or hospital emergency department (ED). During these pain crises, patients sometimes require high doses of opioids for analgesia. Opioid analgesics are fraught with challenges including the development of tolerance, dependence, and opioid-induced hyperalgesia (whereby the use of opioids actually makes patients more sensitive to pain). Finding non-opioid alternatives for intravenous analgesia is problematic based on the limited availability this class of drugs. Ketamine is a potent N-methyl-D-aspartate (NMDA) receptor antagonist that even at low doses has demonstrated efficacy as an adjunct to opioids for acute pain control.

OBJECTIVE:

The investigators will determine the comparative efficacy of low doses of ketamine as an adjunct to opioids versus standard care (opioids alone) for the treatment of acute severe pain in patients with sickle cell related pain crisis.

METHODS:

The investigators propose a double-blinded, randomized, placebo-controlled pilot study to determine the efficacy of ketamine 0.3mg/kg vs. placebo for the treatment of acute pain crisis. The investigators will include all eligible emergency department ≥18 years. The investigators will stratify 42 patients by location, 21 patients per site. Numeric Rating Scale (NRS) will be recorded as a part of the study log at 0, 1, 2 and 3hrs after the study drug administration.

HYPOTHESIS:

The investigators hypothesize that the ketamine will decrease overall pain intensity, visit length of stay, and hospitalizations.

DETAILED DESCRIPTION:
Current treatment standard for acute pain crisis in sickle cell disease (SCD) is largely supportive care: opioid analgesics, hydration, oxygen, and blood transfusion. Sickle cell disease (SCD) is a chronic condition associated with serious and disabling acute consequences such as a vaso-occlusive (VOC) or pain crisis. Uncontrolled pain is the hallmark of a VOC, and often results in acute unscheduled care in the patient's clinic or hospital emergency department (ED). The pain associated with acute VOC in sickle cell disease is caused by the change in the structure of red blood cells. This change leads to microvascular obstruction, a decrease in laminar blood flow, diminished tissue oxygen exchange, and ultimately microenvironmental changes resulting in severe pain.1 During these pain crises, patients sometimes require high doses of opioids for analgesia. Poor pain control, in the setting of high dose opioid administration, is the most common reason for a patient to be hospitalized with acute VOC. Opioid analgesics are fraught with challenges including the development of tolerance, dependence, and opioid-induced hyperalgesia (whereby the use of opioids actually makes patients more sensitive to pain). Finding non-opioid alternatives for intravenous analgesia is problematic based on limited availability and poor side-effect profile. One alternative suggested for use in patients with VOC is ketamine, a potent N-methyl-D-aspartate (NMDA) antagonist.

The current evidence suggests that the counterintuitive effects of opioids are related to activation of NMDA receptors. These effects may be more pronounced in patients with sickle cell disease, as approximately half of these patients have chronic pain and are on long term opioids. The NMDA receptor is activated in response to injury of inflammation, precipitating heightening pain perception, and is therefore an important analgesic target for patients receiving opioids. Ketamine is a potent NMDA receptor antagonist that even at low doses has demonstrated efficacy as an adjunct to opioids for acute pain control. Multiple emergency department studies have shown that low doses of ketamine, <1mg/kg, provides analgesic effects, decreases pain scores, and decreases total opioid use.2-4 While these studies do not focus specifically on adult patients with SCD, ketamine has shown promise in similar pediatric populations. Unfortunately, there are no high-quality studies examining ketamine usage in adult patients with SCD, making highly addictive opioid medications the standard for pain relief during a crisis. The goal of this study is to determine the effectiveness of one non-opioid analgesic, ketamine, in the treatment of acute pain in a vulnerable patient population.

PRIMARY AIM: The investigators will determine the comparative efficacy of low doses of ketamine as an adjunct to opioids versus standard care (opioids alone) for the treatment of acute severe pain in patients with sickle cell related pain crisis. The investigators propose a double-blinded, randomized, placebo-controlled pilot study. The primary outcome will be assessed by patient-reported pain intensity and use of rescue opioid analgesia. Adverse events, length of the encounter, and hospitalization will be evaluated as secondary outcomes. Our central hypothesis is that the ketamine will decrease overall pain intensity, visit length of stay, and hospitalizations. The investigators will enroll patients at both a community hospital emergency department and a tertiary care, academic center. Both locations evaluate and treat patients with acute VOC and will provide an adequate volume for this pilot trial. At the end of this study the investigators expect to determine the effectiveness of ketamine in the treatment of acute pain in patients with SCD presenting after a VOC. Our team is composed of physician-scientists, competent and confident in conducting both clinical and methodological aspects of the trial.

ELIGIBILITY:
Inclusion Criteria:

* All English-speaking adult patients >=18yrs old patients presenting with acute pain crisis

Exclusion Criteria:

* Inability to provide consent,
* Allergy to ketamine
* Pregnant or breastfeeding. W
* Signs and symptoms of intracranial hypertension
* Neurologic deficits
* Headache only
* Temperature >102F
* Sustained blood pressure >=180/110
* Sustained heart rate >130
* Current priapism
* Patients requiring a blood transfusion at the time of acute presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 4 hours
  We anticipate a decrease in numeric pain score after ketamine administration

SECONDARY OUTCOMES:
Emergency department length of stay | 4 hours
  We anticipate a decrease in the LOS in the ED

CONTACTS AND LOCATIONS:
Overall Officials: Taneisha Wison, MD, ScM, Principal Investigator — Brown Emergency Medicine
Locations (2):
- United States (2):
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No
No plan at this time to share IPD with other researchers.